CLINICAL TRIAL: NCT00298571
Title: Cesarean Delivery and Post-operative Pain Management With Local Anesthesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1212
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2006-02

CONDITIONS: Pain, Postoperative
Keywords: Cesarean Delivery; Post-operative; Pain; Local Anesthetic
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Epinephrine

INTERVENTIONS:
Drug: .5% bupivacaine with epinephrine

SUMMARY:
The use of .5% Bupivacaine with epinephrine at the time of skin closure in cesarean deliveries will decrease post-op pain.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL

Title: Cesarean Delivery and Postoperative Pain Management with Local Anesthesia

Investigators: Aaron Deutsch, MD, Principal Investigator Shelly Holmstrom, MD

Abstract:

Pain control has become a more prominent clinical issue. Typically, a patient undergoing a Cesarean delivery is administered spinal anesthesia just prior to the surgery.

Postoperative pain is managed with intravenous (IV) narcotics using a patient controlled anesthesia (PCA) pump device. Once the patient can tolerate oral medications, the PCA pump is discontinued and the patient uses oral narcotic medications for pain control.

Research has shown that injecting a local anesthetic in the subcutaneous tissue along the incision can reduce postoperative pain. The objective of this study is randomly assign patients to receive a local anesthetic or normal saline in the tissues surrounding the incision and to study the amount of pain experienced postoperatively in these groups of patients. Our hypothesis is that the patients receiving the local anesthesia along their incision will have significantly less pain postoperatively and use less narcotic medications.

Objectives:

Primary: To decrease postoperative pain in women undergoing Cesarean delivery Secondary: To decrease narcotic use, potentially decrease hospital length of stay, and increase patient satisfaction

Background, Study Rationale and Significance:

Local anesthesia injected at the incision site fro reduced postoperative pain has been studied in other abdominal surgeries. The research has demonstrated the effectiveness of this technique for reduced postoperative pain. One journal article describes a technique similar to the proposed research project1. However, this article did not show any significant difference in the postoperative pain following bupivacaine or normal saline injection of the skin. The authors' conclusion for this lack of significance was due to their facility's high quality analgesia via supplemental subarachnoid morphine.

Numerous other authors have demonstrated the effectiveness of using local anesthesia at incision sites for reducing pain postoperatively2-4. The proposed research project has the potential to decrease pain postoperatively, decrease hospital length of stay and increase patient satisfaction for one of the most common surgeries in the United States of America.

1. Rajakulendran Y, Chan A. "The Effect of Postoperative Skin Infiltration with Bupivacaine on Postoperative Pain Following Cesarean Section under Spinal Anesthesia." International Journal of Obstetric Anesthesia. Oct 1994;Vol 3(4):199-202
2. Einarsson JI, Sun J, Orav J, Young A. "Local Anesthesia in Laparoscopy: A Randomized Trial." Obstetrics and Gynecology. Dec 2004; 104:1335-9.
3. Lohsiriwat V, Lert-akyamanee N, Rushatamukayanunt W. "Efficacy of Pre-incisional Bupivacaine Infiltration on Postoperative Pain relief after Appendectomy: Prospective Double-Blind Randomized Trial. World Journal of Surgery. 2004 Oct; 28(10):947-50.
4. Khaira HS, Wolf JS Jr. "Intraoperative Local Anesthesia Decreases Postoperative Parental Opioid Requirements fro Transperitoneal Laparoscopic Renal and Adrenal Surgery: A Randomized, Double-blind, Placebo Controlled Investigation. Journal of Urology. 2004 Oct; 172(4 Pt1):1422-6.

Study Population:

Patients currently undergoing a repeat Cesarean delivery with a history of a previous Cesarean delivery through a Pfannenstiel skin incision will be eligible to enroll in this study. All ages and races will be eligible. Exclusion criteria include patients with a primary Cesarean delivery, prior vertical skin incision or an allergy to bupivacaine. The projected sample size required for this study is 100 (50 patients in each arm).

Study Procedures

Research Plan:

This study is a randomized double blind placebo controlled trial. Patients will be randomized to either the bupivacaine or placebo (normal saline) group. An opaque envelope will contain a slip of paper indicating which fluid is to be injected. The anesthesiologist will open the envelope during the surgery and prepare 30 ml of the study drug. The patients will have their incision site injected with either the bupivacaine or normal saline at the completion of the surgery. The patients will be asked to assess their level of pain following the surgery on postoperative days 0, 1, 2 and 3 using a visual analog scale (VAS).

Expected results:

The hypothesis is that the patients receiving the bupivacaine injection will experience significantly less postoperative pain and use significantly less IV and oral narcotic medications.

Human Subject Issues

* there are minimal to no additional risks to the patients in this study. Bupivacaine is a time proven safe drug (barring patient not allergic) and our dose will be far below toxicity levels. There are no social risks or risks of confidentiality as patients will not be personally identified in the study.
* benefits: the benefits to the patient would be a higher satisfaction due to better pain control. Additionally, patients may require less narcotics post-operatively and a potentially shorter hospital stay.
* patient information will be kept track of via name and med rec number for chart review after study completion to assess all data. This info will be limited to only the primary investigators.
* of note the fetus will be delivered prior to the time of anesthetic administration, so they will not be exposed.

Informed Consent Informed consent will be obtained at the time of consent for cesarian delivery. The resident obtaining consent will also obtain the research consent. This will consist of explaining that the patient may receive either a local anesthetic or placebo to help assess better post-op pain control. Possible benefits will be explained along with minimal risks- no more than normal for a cesarian delivery.

The consent process will be available in Spanish and English when applicable.

Statistical Plan

* sample size/power analysis: statistical power for the study to show a statistical difference was calculated to approx 33 patients in each arm- we will extend to 50.
* statistical analysis:

Data Forms and Questionaire (see attached)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women with scheduled cesarean delivery
* able to perform informed consent

Exclusion Criteria:

* Labor
* chronic pain
* allergic to local anesthetic
* unable to perform informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
1. Decreased post-op pain
2. Decreased post-op narcotic use

SECONDARY OUTCOMES:
improved hospital stay satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Holmstrom, MD, Study Director — USF Department OB/Gyn
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States